CLINICAL TRIAL: NCT04480593
Title: The Use of Brazilian Green Propolis Extract (EPP-AF) in Patients Affected by COVID-19: a Randomized, Open and Pilot Clinical Study.
Brief Title: The Use of Brazilian Green Propolis Extract (EPP-AF) in Patients Affected by COVID-19.
Acronym: Bee-Covid
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Marcelo Silveira, Principal Investigator, D'Or Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31099320.6.0000.0048
Record Dates: First submitted 2020-07-12; First posted 2020-07-21 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Propolis; Covid19; SARS-CoV-2; Anti-inflammatory
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: three parallel groups randomly assigned
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the results of interest to the study will not have access to the study steps before the analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): standard care.
  Interventions: Other: Standard care
- EPP-AF 400mg/day (Experimental): Green propolis extract (EPP-AF) at a dose of 400mg / day in addition to the standard treatment.
  Interventions: Drug: Brazilian Green Propolis Extract (EPP-AF)
- EPP-AF 800mg/day (Experimental): Green propolis extract (EPP-AF) at a dose of 800mg / day in addition to the standard treatment.
  Interventions: Drug: Brazilian Green Propolis Extract (EPP-AF)

INTERVENTIONS:
Drug: Brazilian Green Propolis Extract (EPP-AF) — Green propolis extract (EPP-AF) administered orally or via nasoenteral tube.
  Other Names: Standard care
  Arms: EPP-AF 400mg/day; EPP-AF 800mg/day
Other: Standard care — Standard treatment includes, as needed, supplemental oxygen (non-invasive and invasive), antibiotics or antivirals, corticosteroids, vasopressor support, renal replacement therapy and extracorporeal membrane oxygenation (ECMO).
  Arms: Control

SUMMARY:
The COVID-19 pandemic is of grave concern due its impact on human health and on the economy. Propolis, a natural resin produced by bees from plant materials, has anti-inflammatory, immunomodulatory, anti-oxidant properties, and various aspects of the SARS-CoV-2 infection mechanism are potential targets for propolis compounds. Propolis components have inhibitory effects on the ACE2, TMPRSS2 and PAK1 signaling pathways; in addition, antiviral activity has been proven in vitro and in vivo. This is a pilot randomized study that aims to assess the impact of using Brazilian green propolis extract against the deleterious effects of the new coronavirus.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients;
* Positive RT-PCR for SARS-CoV-2;
* 18 Years and older.

Exclusion Criteria:

* Pregnant women;
* People with active cancer;
* Patients undergoing transplantation of solid organs or bone marrow or who use immunosuppressive medications;
* HIV carriers;
* Allergy to propolis or any of its components;
* Bacterial infection at randomization;
* Sepsis or septic shock before randomization;
* Patients unable to use medication orally or via nasoenteral tube;
* Patients with severe chronic liver disease (Child B or C);
* Patients with advanced heart failure;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Composite clinical outcome with oxygen therapy dependency time or hospitalization time | 1-28 days
  Composite clinical outcome with oxygen therapy dependency time (in days) or hospitalization time (in days) after randomization.

SECONDARY OUTCOMES:
Percentage of participants with adverse events during the use of propolis | 1-28 days
  We will evaluate the presence or absence of symptoms related to the use of propolis through a questionnaire.
Rate and severity of acute kidney injury during the study | 1-28 days
  Assess the degree of acute kidney injury according to KDIGO (through serum creatinine or urine output).
Renal replacement therapy. | 1-28 days
  Assess need or not for renal replacement therapy.
Rate of need for vasopressor use | 1-28 days
  Describe the time needed for vasopressors in days after randomization
Need for intensive care unit (ICU) | 1-28 days
  Assess length of stay in the ICU after randomization in days
Intensive care unit (ICU) readmission | 1-28 days
  Rate of readmission to the ICU after randomization
Invasive oxygenation time | 1-28 days
  Assess the need for mechanical ventilation in days after randomization.
Variation of plasma c-reactive protein | 1-7 days
  Evaluate the variation in serum levels of c-reactive protein over the 7 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Silveira, MD, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- Hospital Sao Rafael, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hori JI, Zamboni DS, Carrao DB, Goldman GH, Berretta AA. The Inhibition of Inflammasome by Brazilian Propolis (EPP-AF). Evid Based Complement Alternat Med. 2013;2013:418508. doi: 10.1155/2013/418508. Epub 2013 Apr 16. PMID 23690844
- [Result] Sanders JM, Monogue ML, Jodlowski TZ, Cutrell JB. Pharmacologic Treatments for Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 May 12;323(18):1824-1836. doi: 10.1001/jama.2020.6019. PMID 32282022
- [Result] Maruta H, He H. PAK1-blockers: Potential Therapeutics against COVID-19. Med Drug Discov. 2020 Jun;6:100039. doi: 10.1016/j.medidd.2020.100039. Epub 2020 Apr 19. PMID 32313880
- [Result] Serkedjieva J, Manolova N, Bankova V. Anti-influenza virus effect of some propolis constituents and their analogues (esters of substituted cinnamic acids). J Nat Prod. 1992 Mar;55(3):294-302. doi: 10.1021/np50081a003. PMID 1593279
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Machado JL, Assuncao AK, da Silva MC, Dos Reis AS, Costa GC, Arruda Dde S, Rocha BA, Vaz MM, Paes AM, Guerra RN, Berretta AA, do Nascimento FR. Brazilian green propolis: anti-inflammatory property by an immunomodulatory activity. Evid Based Complement Alternat Med. 2012;2012:157652. doi: 10.1155/2012/157652. Epub 2012 Dec 19. PMID 23320022
- [Result] Mani JS, Johnson JB, Steel JC, Broszczak DA, Neilsen PM, Walsh KB, Naiker M. Natural product-derived phytochemicals as potential agents against coronaviruses: A review. Virus Res. 2020 Jul 15;284:197989. doi: 10.1016/j.virusres.2020.197989. Epub 2020 Apr 30. PMID 32360300
- [Result] Silveira MAD, Teles F, Berretta AA, Sanches TR, Rodrigues CE, Seguro AC, Andrade L. Effects of Brazilian green propolis on proteinuria and renal function in patients with chronic kidney disease: a randomized, double-blind, placebo-controlled trial. BMC Nephrol. 2019 Apr 25;20(1):140. doi: 10.1186/s12882-019-1337-7. PMID 31023272
- [Result] Cusinato DAC, Martinez EZ, Cintra MTC, Filgueira GCO, Berretta AA, Lanchote VL, Coelho EB. Evaluation of potential herbal-drug interactions of a standardized propolis extract (EPP-AF(R)) using an in vivo cocktail approach. J Ethnopharmacol. 2019 Dec 5;245:112174. doi: 10.1016/j.jep.2019.112174. Epub 2019 Aug 20. PMID 31442620